CLINICAL TRIAL: NCT06562751
Title: Developing an Intervention to Help Nurses Improve the Assessment and Care of the Sexual Health Needs of Men With Inflammatory Bowel Disease: a Mixed Methods Study Using Co-production
Brief Title: Developing an Intervention to Help Nurses Improve Sexual Healthcare in Men With Inflammatory Bowel Disease
Acronym: MenSH-IBD
Status: Active, not recruiting | Type: Observational
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of York (Other); York St John University (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: MenSH-IBD
Record Dates: First submitted 2024-07-05; First posted 2024-08-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires; Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Survey 1 (National Health Service Inflammatory Bowel Disease services): A survey designed by the investigators to ascertain current Inflammatory Bowel Disease service provision for sexual healthcare. A representative from each service will complete one online survey that should take approximately 15 minutes to complete.
  Interventions: Other: Questionnaire
- Survey 2 (Inflammatory Bowel Disease nurses survey): A survey designed by the investigators to ascertain current nursing practice for sexual healthcare within Inflammatory Bowel Disease (IBD) services. Registered nurses working with people with IBD will complete one online survey that should take approximately 15 minutes to complete.
  Interventions: Other: Questionnaire
- Survey 3 (men with IBD): A survey designed by the investigators to ascertain the needs of men with Inflammatory Bowel Disease (IBD). Men with a diagnosis of IBD will complete one online survey that should take approximately 15 minutes to complete.
  Interventions: Other: Questionnaire
- Interviews: Men with a diagnosis of Inflammatory Bowel Disease (IBD) and the partners of men with IBD will undertake online, semi-structured interviews that will last no longer than 60 minutes. Participants can be interviewed with their partner or individually. Participants without a partner or whose partner does not wish to be interviewed will be interviewed individually.
  Interventions: Other: Interview
- Focus Groups: Healthcare professionals and appropriate stakeholders (for example charitable organisations) will participate in focus groups. Each focus group will contain 6-8 members. There will be three groups in total.
  Interventions: Other: Focus group
- Co-production workshops: A group of 8-12 inclusive of men with IBD, the partners of men with IBD and healthcare professionals and appropriate stakeholders will participate in three co-production workshops to develop a prototype intervention and logic model to patient benefit.
  Interventions: Other: Workshop

INTERVENTIONS:
Other: Questionnaire — Online questionnaire designed by the investigatory team.
  Groups: Survey 1 (National Health Service Inflammatory Bowel Disease services); Survey 2 (Inflammatory Bowel Disease nurses survey); Survey 3 (men with IBD)
Other: Focus group — Online focus group
  Groups: Focus Groups
Other: Interview — Online semi-structured interview
  Groups: Interviews
Other: Workshop — Online and face to face co-production workshops
  Groups: Co-production workshops

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic, relapsing and remitting disease that can greatly impact health and personal well-being. Sexual health, relationships and intimacy have been raised as key concerns for those living with the disease. Men's sexual health and well-being has been identified as a neglected area. This study will lead to the development of an intervention that will help nurses to improve the assessment and care of the sexual health and well-being needs of men with IBD.

DETAILED DESCRIPTION:
This research aims to develop an intervention to help nurses improve the assessment and care of the sexual health needs of men with Inflammatory Bowel Disease (IBD). This is a long-term digestive condition that is often diagnosed between the ages of 15-30 years. Patients often have bloody diarrhoea, abdominal pain, incontinence, and fatigue.

When severe, the disease can lead to hospital admission and surgery. There is growing recognition that IBD can negatively affect sexual health and impact on patients' relationships and quality of life, but men's needs have been neglected in research. Men report that their sexual health is rarely discussed at National Health Service (NHS) IBD clinic appointments, and specialist information and support are lacking. In this study the investigators will work with men with IBD, the partners of men with IBD, nurses, and other healthcare professionals to develop a nursing intervention that addresses this unmet need through information, assessment, and support.

This study consists of three main parts which have been labelled workstreams. In Workstream One the investigators will identify how the sexual health of men with IBD is currently assessed and cared for in the NHS using three large scale surveys that will include; (1) NHS Trusts (2) Nurses (3) People with IBD.

In Workstream Two the investigators will gather ideas on appropriate ways to improve the healthcare of men with IBD by conducting interviews with men with IBD and partners of men with IBD. The investigators will also conduct focus groups with healthcare professionals to hear their ideas of how services can be improved.

In Workstream Three the investigators will hold a series of workshops with patients and healthcare professionals to develop an intervention and consider how and why it could help patients.

The design of the study has been developed with a patient advisory group and input from IBD health professionals.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of Crohn's Disease, Ulcerative Colitis or IBD-U who identifies as male OR Currently in (or in the last 5 years) an intimate partnership with a person who identifies as male and has a diagnosis for Crohn's Disease, Ulcerative Colitis or IBD-U.

OR An NHS employee whose current employment involves oversight of the delivery and provision of a secondary care IBD patient service within their employing organisation. This may be a healthcare professional or non-clinical manager.

OR A registered nurse who as part of their current role is responsible of the provision of care to patients with IBD.

OR A health professional registered with the GMC, NMC or HCPC whose professional role is considered part of the IBD multidisciplinary team. Currently or previously employed in a role that directly provides care, support or advice to men with a diagnosis of IBD.

OR A representative of a charitable, not-for profit, professional, public or governmental organisation that is engaged with men who suffer from long term conditions or IBD specifically.

Exclusion criteria:

Unable to provide informed consent Less than 18 years old Does not speak English Not able to participate in the research activity (questionnaire, interview, focus group or workshop)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as male
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 792 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Prototype intervention | 18 months
  A prototype intervention to improve the assessment and care of the sexual health needs of men with Inflammatory bowel disease (IBD). The intervention will provide nurses with the improved understanding of the support and knowledge and skills required to effectively assess the sexual health needs of men with Inflammatory Bowel Disease and provide appropriate patient-centred care.

SECONDARY OUTCOMES:
Survey 1 outcomes: | 18 months
  Determine provision of sexual healthcare, assessment and support services to men with IBD in UK National Health Services including whether these differ between male and female patients.
Survey 2 outcome | 18 months
  Facilitators, barriers and confidence of nurses to delivery sexual health assessment, care and advice to male patients.
Survey 3 outcome | 18 months
  Perceived needs, preferences and barriers in regards to sexual health in men with Inflammatory Bowel Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ma, MSc, Principal Investigator — York St John University
Locations (1):
- Sarah Ma, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma S, Forshaw G, Kanaan M, Knapp P, Robinson W, Selinger C, Galdas P. Developing an Intervention to Improve Sexual Health Assessment and Care in Men With Inflammatory Bowel Disease. J Adv Nurs. 2025 Sep 5. doi: 10.1111/jan.70199. Online ahead of print. PMID 40913018

DOCUMENTS (2):
  • Study Protocol (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT06562751/Prot_002.pdf
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT06562751/ICF_001.pdf